CLINICAL TRIAL: NCT02819999
Title: A Study of Rovalpituzumab Tesirine (SC16LD6.5) in the Frontline Treatment of Patients With Extensive Stage Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRX001-004
Record Dates: First submitted 2016-06-27; First posted 2016-06-30 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2019-06

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — rovalpituzumab tesirine; Cisplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Rovalpituzumab Tesirine (Experimental): Rovalpituzumab Tesirine 0.3 mg/kg IV infusion
  Interventions: Drug: Rovalpituzumab Tesirine
- Rovalpituzumab Tesirine followed by Cisplatin, Etoposide (Experimental): Rovalpituzumab Tesirine 0.3 mg/kg IV infusion followed by Cisplatin 80 mg/m2 and Etoposide 100 mg/m2 IV infusion
  Interventions: Drug: Rovalpituzumab Tesirine; Drug: Cisplatin; Drug: Etoposide
- Rovalpituzumab Tesirine with Cisplatin, Etoposide (Experimental): Cisplatin 80 mg/m2 and Etoposide 100 mg/m2 IV infusion and Rovalpituzumab Tesirine 0.1 mg/kg IV infusion
  Interventions: Drug: Rovalpituzumab Tesirine; Drug: Cisplatin; Drug: Etoposide
- Rovalpituzumab Tesirine following Cisplatin, Etoposide (Experimental): Cisplatin 80 mg/m2 and Etoposide 100 mg/m2 IV infusion followed by Rovalpituzumab Tesirine 0.3 mg/kg IV infusion
  Interventions: Drug: Rovalpituzumab Tesirine; Drug: Cisplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Rovalpituzumab Tesirine — Rovalpituzumab tesirine is a DLL3 targeted antibody drug conjugate (ADC).
  Other Names: SC16LD6.5
Drug: Cisplatin
  Arms: Rovalpituzumab Tesirine followed by Cisplatin, Etoposide; Rovalpituzumab Tesirine following Cisplatin, Etoposide; Rovalpituzumab Tesirine with Cisplatin, Etoposide
Drug: Etoposide
  Arms: Rovalpituzumab Tesirine followed by Cisplatin, Etoposide; Rovalpituzumab Tesirine following Cisplatin, Etoposide; Rovalpituzumab Tesirine with Cisplatin, Etoposide

SUMMARY:
The purpose of the study is to test the effect of rovalpituzumab tesirine in the frontline treatment of small cell lung cancer (SCLC).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years with histologically- or cytologically-confirmed, extensive-stage, chemotherapy-naïve SCLC
* DLL3-expressing SCLC based on central immunohistochemistry (IHC) assessment. Positive is defined as staining in ≥75% of tumor cells.
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* Minimum life expectancy of at least 12 weeks.
* Recovery to Grade 1 of any clinically significant toxicity (excluding alopecia) prior to initiation of study drug.
* Satisfactory laboratory parameters within defined parameters (ANC, platelet count, Hb, total bilirubin, ALT, AST and GFR)
* Subjects with a history of CNS metastases must have completed definitive treatment prior to first dose of study treatment, off or on a stable dose of corticosteroids
* Use of effective contraception method during and for 1 year following study drug dosing if female of childbearing potential or sexually active male

Exclusion Criteria:

* Prior systemic chemotherapy, small molecule inhibitors, immune checkpoint inhibitors, other monoclonal antibodies, antibody-drug conjugates, radioimmunoconjugates, T-cell or other cell-based or biologic therapies, or any other anticancer therapy for the treatment of (limited or extensive) SCLC.
* Any significant medical condition, that, in the opinion of the investigator or sponsor, may place the subject at undue risk from the study.
* Documented history of a cerebral vascular, unstable angina, myocardial infarction, or cardiac symptoms consistent with New York Heart Association (NYHA) Class III-IV within 6 months prior to their first dose of study drug.
* Recent or ongoing serious infection.
* Women who are pregnant or breastfeeding.
* History of another invasive malignancy that has not been in remission for at least 3 years. Exceptions: nonmelanoma skin cancer, curatively treated localized prostate cancer, and cervical cancer in situ on biopsy or squamous intraepithelial lesion on PAP smear.
* Prior exposure to a pyrrolobenzodiazepine (PBD)-based drug, or known hypersensitivity to rovalpituzumab tesirine or excipient contained in the drug formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-10; Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT) of rovalpituzumab tesirine when administered as monotherapy, in series or in combination with frontline chemotherapy to subjects with DLL3 expressing extensive-stage small cell lung cancer (SCLC) | within 21 days after first dose of rovalpituzumab tesirine
  For Phase 1a
Treatment emergent adverse events (TEAEs) | through 30 days after last dose of study treatment
  For Phase 1a
Incidence of subjects with CTCAE Grade >2 laboratory abnormalities | through 30 days after last dose of study treatment
  For Phase 1a
Progression-Free Survival (PFS) | 4 years
  For Phase 1b

SECONDARY OUTCOMES:
Best overall response rate | 4 years
Duration of response (DOR) | 4 years
Clinical Benefit Rate (CBR) | 4 years
Overall Survival (OS) | 4 years
Incidence of anti-therapeutic antibodies (ATAs) against rovalpituzumab tesirine | 4 years
Progression-free survival (Phase 1a) | 4 years
Pharmacokinetic parameters: Cmax (Maximum plasma concentration observed ) | 4 years
Pharmacokinetic parameters: AUC0-tau (Area under the plasma concentration-time curve within a dosing interval) | 4 years
Pharmacokinetic parameters: AUC0-∞ (Area under the curve from time 0 extrapolated to infinity) | 4 years
Pharmacokinetic parameters: Tmax (Time of Cmax) | 4 years
Pharmacokinetic parameters: Ctrough (Observed plasma concentrations at trough) | 4 years
Pharmacokinetic parameters: T1/2 (Terminal half-life) | 4 years
Pharmacokinetic parameters: CL (Clearance) | 4 years
Pharmacokinetic parameters: Vss (Volume of distribution at steady state) | 4 years
Incidence of TEAEs | 4 years
  For Phase 1b
Changes in vital signs (Heart Rate) | 4 years
Changes in vital signs (Blood pressure) | 4 years
Changes in vital signs (Temperature) | 4 years
Changes in vital signs (Weight) | 4 years
Changes in vital signs (Respirations) | 4 years
Eastern Cooperative Oncology Group (ECOG) score | 4 years

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of Colorado, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Cancer Institute of Florida, Orlando, Florida
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - Oncology Hematology Care, Cincinnati, Ohio
  - University Hospital of Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Oncology, Fort Worth, Texas
  - Texas Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No